CLINICAL TRIAL: NCT00002022
Title: Treatment Program for Anemia in AIDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R W Johnson Pharmaceutical Research Institute (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 004G; I88-083
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-02

CONDITIONS: HIV Infections; Cytopenias
Keywords: Recombinant Proteins; Drugs, Investigational; Erythropoietin; Acquired Immunodeficiency Syndrome; Anemia; Zidovudine
MeSH Terms: conditions — HIV Infections; Cytopenia; Acquired Immunodeficiency Syndrome; Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The objective of the Eprex (erythropoietin) Treatment Program is to provide erythropoietin for the treatment of anemia in AIDS patients.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Life expectancy < 3 months.
* = or < grade 4 performance score.
* AIDS-related dementia.
* Uncontrolled hypertension.
* Acute symptomatic opportunistic infection or other AIDS-defining illness.

Patients with the following are excluded:

* Life expectancy < 3 months.
* = or < grade 4 performance score.
* AIDS-related dementia.
* Uncontrolled hypertension.
* Acute symptomatic opportunistic infection or other AIDS-defining illness.

Patients must have:

* A clinical diagnosis of AIDS.
* Hematocrit < 30 percent.
* Endogenous serum erythropoietin level = or < 500 U/ml.
* A life expectancy = or > 3 months.
* > Grade 4 performance score.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- R W Johnson Pharmaceutical Research Institute, Raritan, New Jersey, United States